CLINICAL TRIAL: NCT07373145
Title: PRospective Evaluation of Vascular Alterations in CT Angiography After Intervention With Drug-coated Balloon (PREVAIL) Study
Brief Title: Prospective CT Assessment After DCB
Acronym: PREVAIL
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ulsan University Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); KangWon National University Hospital (Other); Korea University Guro Hospital (Other); Sejong General Hospital (Other); Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: H-2404-105-1532; ERP-2024-13777 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2025-08-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: drug coated balloon; CCTA; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with a drug-coated balloon for de novo lesions.: Patients who underwent DCB within 3 months after CCTA and whose clinical presentation remained largely unchanged from the time of CCTA.

SUMMARY:
This prospective, multicenter observational cohort study aims to investigate changes in target lesion hemodynamic parameters, diameter stenosis, plaque characteristics of CCTA before and after the DCB procedure and evaluate their association with clinical outcomes.

DETAILED DESCRIPTION:
This prospective, multicenter observational cohort study will include patients with coronary artery disease who underwent drug-coated balloon (DCB) treatment and had coronary computed tomography angiography (CCTA) performed at baseline. Follow-up CCTA will be conducted two years after the index DCB procedure. The study aims to evaluate changes in target lesion hemodynamic parameters, diameter stenosis, and plaque characteristics on CCTA before and after DCB treatment, and to assess their association with subsequent clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Age ≥ 19
* Patients who took CCTA and were found to have coronary artery disease requiring reperfusion
* Patients who underwent DCB within 3 months after CCTA and whose clinical presentation remained largely unchanged from the time of CCTA.
* The target lesion is a de novo lesion with a vessel diameter between 2.25mm and 3.00mm
* Patients deemed suitable for coronary intervention using drug-coated balloon by clinical assessment
* Patients who have been adequately informed about this study and have voluntarily provided written consent to participate.

Exclusion Criteria:

* The target lesion is an in-stent restenosis lesion
* Patient requiring emergency salvage stenting in target lesion
* Patients with a stent previously implanted in the same vessel
* Lesions involving chronic total occlusion or prior coronary artery bypass grafting (CABG).
* Patients with eGFR (estimated glomerular filtration rate) < 45 ml/min/1.73mm2
* Patients with coronary artery calcium score ≥ 1000 as determined by CCTA
* Patients with an expected survival of less than 5 years
* Pregnant or breastfeeding patients
* Patients deemed inappropriate to participate in this study based on the judgment of study investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who took coronary computed tomography angiography (CCTA) and received drug-coated balloon (DCB) treatment for coronary artery disease
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ΔFFR CT before and after DCB procedure | From baseline CCTA to follow-up CCTA performed 2 years after the index PCI

SECONDARY OUTCOMES:
Changes in plaque characteristics before and after DCB procedure | From baseline CCTA to follow-up CCTA performed 2 years after the index PCI
Changes in diameter stenosis before and after DCB procedure | From baseline CCTA to follow-up CCTA performed 2 years after the index PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The sharing plan will be decided by the study committee.